CLINICAL TRIAL: NCT00736515
Title: Phase 4 Study of Comparison of Combination Therapy of Gliclazide MR and Basal Insulin With Pre-mix Insulin Monotherapy for the Patients With Type 2 Diabetes Mellitus
Brief Title: Study of Combination Therapy of Gliclazide MR and Basal Insulin Versus Insulin Monotherapy to Treat Type 2 Diabetes
Acronym: CODMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Servier (Tianjin) Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC4-5702-205-CHN
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes
Keywords: combination therapy,monotherapy,gliclazide MR,insulin,CGMS
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination therapy (Experimental): The subjects allocated into this arm will receive the combination therapy of oral administration of 60~120mg Gliclazide MR (Diamicron MR) and subcutaneous injection of basal insulin (Insulin Glargine Injection, Lantus) once daily for 3 months
  Interventions: Drug: Gliclazide MR and Insulin Glargine Injection
- monotherapy (Active Comparator): The patients allocated into this arm will receive the monotherapy of subcutaneous injection of premixed insulin (Biosynthetic Human Insulin Injection, Novolin 30R) twice daily for 3 months.
  Interventions: Drug: Biosynthetic Human Insulin Injection

INTERVENTIONS:
Drug: Gliclazide MR and Insulin Glargine Injection — Combination therapy of oral administration of 60-120mg Gliclazide Modified Release Tablet once daily before breakfast and subcutaneous injection of Insulin Glargine Injection once daily before dinner (initial dosage 0.2U/KG/D) for 3 months
  Other Names: Brand Name: Diamicron MR and Lantus
  Arms: Combination therapy
Drug: Biosynthetic Human Insulin Injection — Monotherapy of subcutaneous injection of Biosynthetic Human Insulin Injection twice daily (before breakfast and before dinner) (initial dosage 0.4-0.6U/KG/D) for 3 months
  Other Names: Brand Name: Novolin 30R
  Arms: monotherapy

SUMMARY:
In recent years, with the further research of the pathogenesis of diabetes mellitus and the mechanism of oral antidiabetes drugs, the early combination therapy of oral antidiabetes drugs and insulin is getting paid more and more attention. A lot of studies have confirmed that Gliclazide MRs have excellent reducing blood glucose efficacy and vascular protection. Based on these theory and practice, this study is designed to demonstrate whether the combination therapy of Gliclazide MR and basal insulin can control the blood glycemia effectively and reduce the dosage of insulin and the hypoglycemia events compared to the premix insulin monotherapy.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Male or female with type 2 diabetes mellitus
2. 35 years old≤age≤65 years old
3. 19kg/m2≤BMI≤32kg/m2
4. Uncontrolled blood glycemia (FPG≥7.0mmol/L and 7.5%<HbA1c≤10%) after oral antidiabetes drugs treatment for more than 3 months
5. Treated by diet controlling, 1 secretagogue agent and another oral antidiabetes drug, with the daily dosage of the secretagogue agent not more than 50% of its maximum
6. Not participated in other clinical studies within the past 3 months
7. Well know this study and sign the informed consent form

Exclusion criteria:

1. Unable to sign the informed consent form
2. Treated by insulin, even transient usage within the past 1 year
3. Type 1 diabetes mellitus
4. Abnormal condition of gastrointestinal tract against the absorption of oral drugs
5. Insufficient of liver and kidney function: ALT≥2.5 times of the upper limit of the normal value range and serum creatinine≥the upper limit of the normal value range
6. Encountered the cardiovascular events such as the angina pectoris, myocardial infarction, severe ventricular arrhythmia, cerebral hemorrhage, cerebral infarction, heart failure ect. within the past half year
7. Usage of the other hormone medicines such as cortical hormone, immunosuppressive agents or cytotoxic drugs within the past 2 months
8. psychotic
9. Allergic history to sulfonylurea drugs
10. Diabetic coma or diabetic ketoacidosis
11. In use of the miconazole
12. Pregnancy or breeding women

Primary endpoint:

Decreasing value of FPG and HbA1c, Dosage of the insulin, Control rate of FPG

Second Endpoints:

1. MBG, SDBG, MAGE and MODD in the 48th CGMS
2. Incidence of hypoglycemia and severe hypoglycemia
3. Weight change

ELIGIBILITY:
Inclusion criteria:

1. Male or female with type 2 diabetes mellitus
2. 35 years old≤age≤65 years old
3. 19kg/m2≤BMI≤32kg/m2
4. Uncontrolled blood glycemia (FPG≥7.0mmol/L and 7.5%<HbA1c≤10%) after oral antidiabetes drugs treatment for more than 3 months
5. Treated by diet controlling, 1 secretagogue agent and another oral antidiabetes drug, with the daily dosage of the secretagogue agent not more than 50% of its maximum
6. Not participated in other clinical studies within the past 3 months
7. Well know this study and sign the informed consent form

Exclusion criteria:

1. Unable to sign the informed consent form
2. Treated by insulin, even transient usage within the past 1 year
3. Type 1 diabetes mellitus
4. Abnormal condition of gastrointestinal tract against the absorption of oral drugs
5. Insufficient of liver and kidney function: ALT≥2.5 times of the upper limit of the normal value range and serum creatinine≥the upper limit of the normal value range
6. Encountered the cardiovascular events such as the angina pectoris, myocardial infarction, severe ventricular arrhythmia, cerebral hemorrhage, cerebral infarction, heart failure ect. within the past half year
7. Usage of the other hormone medicines such as cortical hormone, immunosuppressive agents or cytotoxic drugs within the past 2 months
8. psychotic
9. Allergic history to sulfonylurea drugs
10. Diabetic coma or diabetic ketoacidosis
11. In use of the miconazole
12. Pregnancy or breeding women

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Decreasing value of FPG and HbA1c, dosage of insulin and control rate of FPG | 3 months

SECONDARY OUTCOMES:
MBG, SDBG, MAGE and MODD in the 48th CGMS | 3 months
Incidence of hypoglycemia and severe hypoglycemia | 3 months
Weight change | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, MD, PHD, Principal Investigator — Shanghai Sixth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine; Jian Zhou, MD, PHD, Study Director — Shanghai Sixth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine; Yuqian Bao, MD, PHD, Study Director — Shanghai Sixth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine; Huazhang Yang, MD, PHD, Study Director — Guangdong Provincial People's Hospital; Jian Kuang, MD, PHD, Study Director — Guangdong Provincial People's Hospital; Hongmei Chen, MD, Study Director — Guangdong Provincial People's Hospital; Haoming Tian, MD, Study Director — West China Hospital; Hong Li, MD, Study Director — SIR RUN RUN SHAW Hospital Affiliated to Zhejiang University School of Medicine; Fenping Zheng, MD, Study Director — SIR RUN RUN SHAW Hospital Affiliated to Zhejiang University School of Medicine; Qiang Li, MD, Study Director — The Second Affiliated Hospital of Harbin Medical University; Xiaohui Guo, MD, PHD, Study Director — Peking University First Hospital; Ying Gao, MD, PHD, Study Director — Peking University First Hospital; Muxun Zhang, MD, Study Director — Tongji Hospital; Lixin Guo, MD, PHD, Study Director — Beijing Hospital; Yan Ren, MD, PHD, Study Director — West China Hospital
Locations (8):
- China (8):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Shanghai Sixth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - SIR RUN RUN SHAW Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Janka HU, Plewe G, Riddle MC, Kliebe-Frisch C, Schweitzer MA, Yki-Jarvinen H. Comparison of basal insulin added to oral agents versus twice-daily premixed insulin as initial insulin therapy for type 2 diabetes. Diabetes Care. 2005 Feb;28(2):254-9. doi: 10.2337/diacare.28.2.254. PMID 15677775
- [Result] Zhou J, Zheng F, Guo X, Yang H, Zhang M, Tian H, Guo L, Li Q, Mo Y, Jia W. Glargine insulin/gliclazide MR combination therapy is more effective than premixed insulin monotherapy in Chinese patients with type 2 diabetes inadequately controlled on oral antidiabetic drugs. Diabetes Metab Res Rev. 2015 Oct;31(7):725-33. doi: 10.1002/dmrr.2661. Epub 2015 Jun 16. PMID 25952634